CLINICAL TRIAL: NCT00586040
Title: Photochemical Tissue Bonding (PTB) for Excisional Wound Healing
Brief Title: Photochemical Tissue Bonding
Acronym: PTB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Irene E. Kochevar, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006p001528
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma; Atypical Nevus
Keywords: skin cancer; skin excision; laser; superficial sutures; wound healing
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Dysplastic Nevus Syndrome; Skin Neoplasms | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): superficial closure with PTB
  Interventions: Procedure: tissue bonding
- 2 (Active Comparator): superficial sutures
  Interventions: Procedure: sutures

INTERVENTIONS:
Procedure: tissue bonding — application of rose bengal and treatment with green light
  Arms: 1
Procedure: sutures — interrupted superficial sutures
  Arms: 2

SUMMARY:
The broad aim of this study is to evaluate the efficacy of photochemical tissue bonding (PTB) for the closure of skin excisions. We will test the hypothesis that full thickness skin excisions treated with PTB can heal with less scarring than those treated with the conventional suture closure method.

DETAILED DESCRIPTION:
Hypertrophic scarring is a frequent endpoint after traditional surgical excision of skin cancers of the chest. These scars create significant long-term morbidity to the patient. There is a clinical need for an alternative treatment that would reduce factors associated with hypertrophic and possibly keloid scar formation by providing minimal tension, low infection risk and an absence of foreign body material. This would result in a normal appearing and healed scar without associated patient morbidity. Photochemical tissue bonding may provide this alternate treatment. PTB differs from sutures by continuously joining the tissue surfaces on a molecular level rather than only at discrete suture points. In addition, PTB does not incite foreign body reactions nor create tissue injury during passage of the needle and tying a knot, injuries that may initiate scarring.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology confirmed basal cell carcinoma or well-differentiated squamous cell carcinoma without subcutaneous fat invasion on the chest, arm or abdomen or a diagnosis of atypical or dysplastic nevi on the chest, arm or abdomen.
* Able to follow involved post-operative care instructions
* Able to comply with study requirements
* Age 20-60 years

Exclusion Criteria:

History of underlying photosensitivity condition Skin phototypes V-VI Use of photosensitizing medication History of Accutane use within the past 12 months History of underlying bleeding disorder or use of anticoagulant (e.g. coumadin) Active smoker Known pregnancy or lactating mother Allergies or reactions to lidocaine or epinephrine Underlying immunodeficiency Inability to comply with study requirements Pacemaker or defibrillator in place

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
scar appearance | 6 months

SECONDARY OUTCOMES:
patient satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Irene E Kochevar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tsao S, Yao M, Tsao H, Henry FP, Zhao Y, Kochevar JJ, Redmond RW, Kochevar IE. Light-activated tissue bonding for excisional wound closure: a split-lesion clinical trial. Br J Dermatol. 2012 Mar;166(3):555-63. doi: 10.1111/j.1365-2133.2011.10710.x. Epub 2012 Jan 19. PMID 22032650
- See also: Wellman Center for Photomedicine — http://www.massgeneral.org/wellman/
- See also: Department of Dermatology, Massachusetts General Hospital — http://www.mgh.harvard.edu/mghdermatology/
- See also: Irene E Kochevar — http://www.massgeneral.org/wellman/people/ikochevar.asp